CLINICAL TRIAL: NCT02180516
Title: Safety and Efficacy of Meloxicam (MOBIC) Compared to Other NSAIDs in Approved Therapeutic Dosages and Routes of Administration in an Observational Cohort Study of Patients With Rheumatoid Arthritis, Osteoarthritis, Lumbago, Scapulohumeral Periarthritis, Neck, Shoulder and Arm Syndrome
Brief Title: Safety and Efficacy of Meloxicam Compared to Other Nonsteroidal Antiinflammatory Drugs (NSAIDs) in an Observational Cohort Study of Patients With Rheumatoid Arthritis, Osteoarthritis, Lumbago, Scapulohumeral Periarthritis, Neck, Shoulder and Arm Syndrome
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 107.246
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Meloxicam; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Meloxicam
  Interventions: Drug: Meloxicam
- Other NSAIDs
  Interventions: Drug: Other Non Steroidal Anti-Inflammatory Drugs (NSAIDs) except etodolac

INTERVENTIONS:
Drug: Meloxicam
  Groups: Meloxicam
Drug: Other Non Steroidal Anti-Inflammatory Drugs (NSAIDs) except etodolac
  Groups: Other NSAIDs

SUMMARY:
Study to assess the safety profile of meloxicam by comparing incidence of gastrointestinal adverse events of meloxicam with that of NSAID in the routine daily therapeutic situation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Indications according to the package insert of the prescribed NSAID

Exclusion Criteria:

* There is no exclusion criterion, because this Post Marketing Study is an observational study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from hospitals or general practioners (Internal Medicine, Orthopedics)
Sampling Method: Non-Probability Sample
Enrollment: 9984 (Actual)
Dates: Start 2001-10; Primary Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Incidence for adverse event of gastrointestinal disorder | up to 6 months

SECONDARY OUTCOMES:
Incidence for adverse drug reaction of gastrointestinal disorder | up to 6 months
Incidence of adverse events | up to 6 months
Incidence of adverse drug reactions | up to 6 months
Incidence of serious adverse events | up to 6 months
Incidence for adverse events Perforation, Ulcer and Bleeding (PUB) in the upper gastrointestinal tract | up to 6 months